CLINICAL TRIAL: NCT00000558
Title: Prevention of Events With Angiotensin-Converting Enzyme Inhibitor Therapy (PEACE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 102
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia | interventions — Angiotensin-Converting Enzyme Inhibitors

INTERVENTIONS:
Drug: angiotensin-converting enzyme inhibitors

SUMMARY:
To determine whether the addition of angiotensin converting enzyme (ACE) inhibitor to standard therapy in patients with known coronary artery disease and preserved left ventricular function will prevent cardiovascular mortality and reduce the risk of myocardial infarction.

DETAILED DESCRIPTION:
BACKGROUND:

Individuals with coronary artery disease are at heightened risk for major cardiovascular events. With current advances, a larger segment of our population is manifesting coronary artery disease at a more advanced age. The majority of these individuals have preserved left ventricular function. Prior studies with converting enzyme inhibitor (CEI) therapy in patients with depressed ejection fraction have demonstrated that their long-term administration leads to improved survival and reduced risk of myocardial infarction over and above conventional therapy. There is sufficient rationale and experience to indicate that these benefits will apply to the larger group of individuals with coronary artery disease and preserved left ventricular function and therefore have even broader public health implications. A definitive trial is needed to assess the capacity of CEI therapy to prevent mortality and reduce the risk of myocardial infarction in patients with coronary disease and preserved left ventricular function.

The initiative was proposed by the former Clinical Trials Branch staff and given concept clearance at the May 1994 National Heart, Lung, and Blood Advisory Council. The Request for Proposals was released in October 1994.

DESIGN NARRATIVE:

A multicenter, randomized clinical trial. There are approximately 180 centers in the United States, Canada, Puerto Rico, and Italy. Patients are randomly assigned to treatment groups in which the addition of the angiotensin-converting enzyme (ACE) inhibitor trandolapril is compared to standard therapy. The primary endpoint includes a reduction in the incidence of cardiovascular death, nonfatal myocardial infarction, or the need for coronary revascularization (PTCA or CABG) in coronary artery disease patients with left ventricular ejection fraction of 40 percent or more. Secondary endpoints include the incidence of hospitalization for the management of either unstable angina, congestive heart failure, stroke, or cardiac arrhythmia. Recruitment started in November 1996 and ended in June 2000 with a minimum follow-up of five years.

ELIGIBILITY:
Men and women patients at least 50 years of age with coronary heart disease documented by angiography and a left ventricular ejection fraction of 40 percent or more.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fowler — George Washington University Biostatistics Center

REFERENCES:
- [Background] Pfeffer MA, Domanski M, Rosenberg Y, Verter J, Geller N, Albert P, Hsia J, Braunwald E. Prevention of events with angiotensin-converting enzyme inhibition (the PEACE study design). Prevention of Events with Angiotensin-Converting Enzyme Inhibition. Am J Cardiol. 1998 Aug 6;82(3A):25H-30H. doi: 10.1016/s0002-9149(98)00488-3. PMID 9719019
- [Background] Pfeffer MA, Domanski M, Verter J, Dunlap M, Flaker GC, Gersh B, Hsia J, Goldberg AD, Limacher MC, Maggioni AP, Rosenberg Y, Rouleau JL, Warnica JW, Wasserman AG, Braunwald E; PEACE Investigators. The continuation of the Prevention of Events With Angiotensin-Converting Enzyme Inhibition (PEACE) Trial. Am Heart J. 2001 Sep;142(3):375-7. doi: 10.1067/mhj.2001.117603. No abstract available. PMID 11526345
- [Background] Braunwald E, Domanski MJ, Fowler SE, Geller NL, Gersh BJ, Hsia J, Pfeffer MA, Rice MM, Rosenberg YD, Rouleau JL; PEACE Trial Investigators. Angiotensin-converting-enzyme inhibition in stable coronary artery disease. N Engl J Med. 2004 Nov 11;351(20):2058-68. doi: 10.1056/NEJMoa042739. Epub 2004 Nov 7. PMID 15531767
- [Derived] Ma T, Zhao J, Yan Y, Liu J, Zang J, Zhang Y, Ruan K, Xu H, He W. Plasma osteoprotegerin predicts adverse cardiovascular events in stable coronary artery disease: the PEACE trial. Front Cardiovasc Med. 2023 Jun 14;10:1178153. doi: 10.3389/fcvm.2023.1178153. eCollection 2023. PMID 37388640
- [Derived] Lachin JM, Bebu I. Application of the Wei-Lachin multivariate one-directional test to multiple event-time outcomes. Clin Trials. 2015 Dec;12(6):627-33. doi: 10.1177/1740774515601027. Epub 2015 Sep 2. PMID 26336199
- [Derived] Udell JA, Morrow DA, Jarolim P, Sloan S, Hoffman EB, O'Donnell TF, Vora AN, Omland T, Solomon SD, Pfeffer MA, Braunwald E, Sabatine MS. Fibroblast growth factor-23, cardiovascular prognosis, and benefit of angiotensin-converting enzyme inhibition in stable ischemic heart disease. J Am Coll Cardiol. 2014 Jun 10;63(22):2421-8. doi: 10.1016/j.jacc.2014.03.026. Epub 2014 Apr 9. PMID 24727254
- [Derived] Omland T, Pfeffer MA, Solomon SD, de Lemos JA, Rosjo H, Saltyte Benth J, Maggioni A, Domanski MJ, Rouleau JL, Sabatine MS, Braunwald E; PEACE Investigators. Prognostic value of cardiac troponin I measured with a highly sensitive assay in patients with stable coronary artery disease. J Am Coll Cardiol. 2013 Mar 26;61(12):1240-9. doi: 10.1016/j.jacc.2012.12.026. Epub 2013 Feb 13. PMID 23414791
- [Derived] Solomon SD, Lin J, Solomon CG, Jablonski KA, Rice MM, Steffes M, Domanski M, Hsia J, Gersh BJ, Arnold JM, Rouleau J, Braunwald E, Pfeffer MA; Prevention of Events With ACE Inhibition (PEACE) Investigators. Influence of albuminuria on cardiovascular risk in patients with stable coronary artery disease. Circulation. 2007 Dec 4;116(23):2687-93. doi: 10.1161/CIRCULATIONAHA.107.723270. Epub 2007 Nov 19. PMID 18025537
- [Derived] Solomon SD, Rice MM, A Jablonski K, Jose P, Domanski M, Sabatine M, Gersh BJ, Rouleau J, Pfeffer MA, Braunwald E; Prevention of Events with ACE inhibition (PEACE) Investigators. Renal function and effectiveness of angiotensin-converting enzyme inhibitor therapy in patients with chronic stable coronary disease in the Prevention of Events with ACE inhibition (PEACE) trial. Circulation. 2006 Jul 4;114(1):26-31. doi: 10.1161/CIRCULATIONAHA.105.592733. Epub 2006 Jun 26. PMID 16801465
- See also: Related Info — http://www.bsc.gwu.edu/peace/
- Available data/document: Individual Participant Data Set: PEACE — http://biolincc.nhlbi.nih.gov/studies/peace/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/peace/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/peace/